CLINICAL TRIAL: NCT05758025
Title: Dissection of Thyroid and Central Lymph Nodes Based on "Layer of Thymus-blood Vessel-inferior Parathyroid Gland" Complex for Preserving the Inferior Parathyroids
Brief Title: A New Surgical Strategy to Protect the Inferior Parathyroid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0077
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection based on "thymus-vascular-inferior parathyroid" complex (Experimental)
  Interventions: Procedure: Resection based on "thymus-vascular-inferior parathyroid" complex
- Traditional thyroidectomy method (No Intervention)

INTERVENTIONS:
Procedure: Resection based on "thymus-vascular-inferior parathyroid" complex — Before clearing the central lymph nodes, looking for the thyro-thymic ligament first, looking for the inferior parathyroid along the thyro-thymic ligament. Dissect and leave the "thymus-vascular-inferior parathyroid" complex laterally; the inner side of this layer is the tissue of the central area. Then remove the central lymph nodes. Check for parathyroids in the removed specimen, transplant the parathyroids which are removed by accident.
  Arms: Resection based on "thymus-vascular-inferior parathyroid" complex

SUMMARY:
The incidence of temporary hypoparathyroidism after thyroid surgery is 14%-60%, and the incidence of permanent hypoparathyroidism is 4%-11%. The protection of parathyroids has always been the focus and difficulty of thyroid surgery. The anatomical position of the superior parathyroids is relatively fixed, and can be preserved in situ easily; while the anatomical position of inferior parathyroids varies greatly between patients. It is always difficult to look for, identify, and protect them. Concepts such as thyro-thymic ligament and "thymus-vascular-inferior parathyroid plane" were raised to help identify the inferior parathyroids. We found that this surgical strategy can protect inferior parathyroids in situ effectively in our retrospective studies. Thus, we are going to carry out a prospective study to compare the new method and the traditional method of thyroidectomy, to see if more inferior parathyroids can be protected in situ through the new surgical strategy.

ELIGIBILITY:
Inclusion Criteria:

* initial thyroid surgery; thyroidectomy with/without central lymph node dissection

Exclusion Criteria:

* coexisting parathyroid disease; need lateral neck dissection; history of radio-iodine ablation treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Postoperative day 1
  the incidence of hypothyroidism

SECONDARY OUTCOMES:
Secondary outcome | Postoperative day 1
  the incidence of parathyroid hormone reduced greater than 50% than parathyroid hormone level before surgery

OTHER OUTCOMES:
Other outcome | 3 weeks after surgery, then every 3 month during the first year after surgery until 12 months after surgery
  time to recover from hypoparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Qunzi Zhao, M.D., Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, ZJ, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang JB, Wu K, Shi LH, Sun YY, Li FB, Xie L. In situ preservation of the inferior parathyroid gland during central neck dissection for papillary thyroid carcinoma. Br J Surg. 2017 Oct;104(11):1514-1522. doi: 10.1002/bjs.10581. Epub 2017 Aug 7. PMID 28782797